CLINICAL TRIAL: NCT06158620
Title: Intra-nasal Ketorolac Versus Oral Diclofenac for Acute Ureteral Stent-associated Pain Following Ureteroscopy for Stone Disease
Brief Title: Intra-nasal Ketorolac for Acute Ureteral Stent-associated Pain Following Ureteroscopy for Stone Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: assertio Therapeutics, Inc (Unknown)
Responsible Party: Principal Investigator, Brett Johnson, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0775
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Pain; Urolithiasis; Ureter Calculi; Stent Complication
MeSH Terms: conditions — Pain, Postoperative; Urolithiasis | interventions — Ketorolac; Diclofenac

STUDY DESIGN:
Intervention Model Description: Phase I will consist of a single-arm open label pilot study. Prior to the initiation of a large-scale randomized trial, we propose a single-arm open label pilot study to evaluate the feasibility, practicality, and qualitative outcomes of utilizing intra-nasal ketorolac in patients with indwelling ureteral stents. We seek to enroll 20 patients for the initial pilot.
  Phase II will consist of a randomized trial comparing intranasal ketorolac to Diclofenac, a commonly used oral NSAID. , Diclofenac potassium. Following ureteroscopy and stent placement, patients will receive standard of care medications to mitigate post operative pain and stent discomfort, and will be randomized to receive either as needed intra-nasal ketorolac or oral diclofenac. We seek to enroll and randomize 60 patients in a 1:1 fashion. Analysis will be intention to treat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sprix (Experimental): Phase I will consist of a single-arm open label pilot study. Prior to the initiation of a large-scale randomized trial, we propose a single-arm open label pilot study to evaluate the feasibility, practicality, and qualitative outcomes of utilizing intra-nasal ketorolac in patients with indwelling ureteral stents. We seek to enroll 20 patients for the initial pilot.
  Phase II will consist of a randomized trial comparing intranasal ketorolac to Diclofenac, a commonly used oral NSAID. , Diclofenac potassium. Following ureteroscopy and stent placement, patients will receive standard of care medications to mitigate post operative pain and stent discomfort, and will be randomized to receive either as needed intra-nasal ketorolac or oral diclofenac. We seek to enroll and randomize 60 patients in a 1:1 fashion. Analysis will be intention to treat.
  Interventions: Drug: intra-nasal ketorolac
- Diclofenac (Active Comparator): Phase II will consist of a randomized trial comparing intranasal ketorolac to Diclofenac, a commonly used oral NSAID. , Diclofenac potassium. Following ureteroscopy and stent placement, patients will receive standard of care medications to mitigate post operative pain and stent discomfort, and will be randomized to receive either as needed intra-nasal ketorolac or oral diclofenac. We seek to enroll and randomize 60 patients in a 1:1 fashion. Analysis will be intention to treat.
  Interventions: Drug: oral diclofenac

INTERVENTIONS:
Drug: intra-nasal ketorolac — Experimental group receiving intra-nasal ketorolac for management of post-operative pain following ureteroscopy for kidney stone, and associated ureter stent discomfort.
  Other Names: Sprix
  Arms: Sprix
Drug: oral diclofenac — Control group to receive oral diclofenac, which is a comparable medication to intra-nasal ketorolac.
  Arms: Diclofenac

SUMMARY:
Objective: To improve quality-of-life and health care delivery to patients receiving ureteral stents.

Specific Aims: Evaluate the feasibility, practicality, and qualitative outcomes of utilizing intra-nasal ketorolac in patients with indwelling ureteral stents (Phase I), followed by a randomized trial comparing two non-steroidal anti-inflammatory drugs, intra-nasal Ketorolac versus oral Diclofenac.

Hypotheses: Due to its favorable pharmacokinetics in relieving acute pain, investigators expect improved pain scores and a lower rate of unplanned clinical encounters in patients receiving intra-nasal ketorolac compared to those taking oral diclofenac following ureteroscopic surgery for urolithiasis.

Study Rationale: Following ureteroscopic management of urolithiasis, patient with indwelling ureter stents have higher levels of discomfort compared to those without a ureter stent. Prior studies showed that intramuscular Ketorolac at time of ureter stent removal decreased the incidence of unplanned clinical encounters. Furthermore, onset of analgesic effect by intra-nasal ketorolac is faster than its oral form, and similar its intramuscular and intravenous counterparts.

DETAILED DESCRIPTION:
Urinary stone disease (USD) leads to pain, diminished quality of life, missed work and school, chronic kidney disease, and renal failure.1-5 The prevalence of kidney stone disease in adults has risen to almost 9% as of 2010 in the United States (US). The 5-year recurrence rate without treatment is 53%.6,7 Increasing utilization of a ureteroscopic approach to treat urolithiasis has led to an increased proportion of stone patients undergoing ureteral stent placement.

In the US, approximately 90% of patients receive a ureteral stent following ureteroscopy. Some patients that undergo ureteral stent placement experience significant and debilitating symptoms of urinary urgency, frequency, suprapubic and flank pain, and incontinence. Treatment of these symptoms has historically relied heavily on opioid pain medications. However, recent emphasis on risk associated with opioid medications has reduced their use, and paved the way for alternative approaches. As such, non-steroidal anti-inflammatory drugs (NSAIDs) have become an integral part of multimodal techniques at mitigating post operative pain and associated ureter stent discomfort.

Ketorolac, an NSAID, can be used in the management of acute pain related to ureteral obstruction, renal colic, and indwelling ureter stent. There are four available formulations of ketorolac: oral, intra-muscular (IM), intra-nasal (IN), and intravenous (IV). Non-oral formulations are known to have faster onset of action and an earlier peak analgesic effect.8 As opposed to injectable (IM or IV) ketorolac that needs to be administered by a clinical provider, IN ketorolac may conveniently be self-administered.9 Furthermore, the favorable pharmacokinetics of IN ketorolac allow for its significant efficacy in providing timely pain relief without the need of opioid medications. However, one of the significant barriers of intra-nasal ketorolac is the cost. An intra-nasal course can cause upwards of $1500 compared to $20 of oral ketorolac.

Ketorolac prevents unplanned renal colic-related clinical encounters post stent removal.10 Study team recently published the study team's results from a randomized trial comparing intramuscular injection of ketorolac to placebo at the time ureteral stent removal reduced the incidence of unplanned clinic returns or emergency room visits. While this trial was aimed at the small number of patients that develop severe ureteral colic following stent removal, investigators feel ketorolac's strong anti-inflammatory properties can be leveraged to mitigate acute indwelling ureteral stent symptoms.

While it is not feasible to treat every stent patient empirically with IN ketorolac, there may be an identifiable subset of patients that may benefit from this formulation. Its favorable pharmacokinetics allow for its significant efficacy in providing timely pain relief without the need of opioid medications. This makes IN ketorolac an intriguing option that may decrease unplanned clinical encounters related to indwelling ureter stent discomfort. Especially when the cost of a post-operative emergency room visits which can include laboratory testing, computed tomography, IV medication and possible admission can dwarf the cost of IN ketorolac.

Furthermore, a recent qualitative analysis published by Harper et al in the in the STudy to Enhance uNderstanding of sTent-associated Symptoms (STENTS) study reveal a highly variable patient experience with stents.11 For some, the negative experience of the stent can be life altering. Therefore, there is a critical need to improve the pain and quality of life of those requiring ureteral stenting. Ideally, this can be done in a directed way to offer more relief to those patients most at risk for severe symptoms.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* English-speaking
* Candidate for unilateral ureteroscopy for treatment of urolithiasis
* Surgical plan includes placement of a ureteral stent

Exclusion Criteria:

* Pregnant/nursing, prisoners, cognitively impaired
* Solitary kidney
* Stone in transplant kidney
* Anatomic abnormalities (i.e., ureteral stricture, infundibular stenosis, uretero-pelvic junction obstruction, horseshoe kidney, duplicated system)
* History of ureteral reconstruction
* History of nephrocalcinosis, medullary sponge kidney, cystinuria
* Immobility or relative immobility
* Planned staged ureteroscopy
* History of ureteral stent complication or poor tolerance or a ureteral stent
* Urinary tract infection or sepsis
* Current anticoagulation use (81 mg Aspirin permissible)
* NSAID contraindication (acute renal failure or chronic kidney disease, bleeding disorders, allergic reaction to NSAIDs, ulcer disease, auto-immune disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores as measured by USSQ Pain Survey | Baseline (before surgery in the pre-operative setting -Day 0), the day of ureter stent removal (Post-operative day 5 through 10)
  Associated pain burden will be measured using standardized Ureteral Stent Symptom Questionnaire (USSQ) Pain Survey. Possible scores range from 0-10, where lower scores indicate better outcome.
Change in pain scores as measured by PROMIS questionnaire | Baseline (before surgery in the pre-operative setting -Day 0), the day of ureter stent removal (Post-operative day 5 through 10)
  Associated pain burden will be measured using standardized Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity and Interference questionnaire. Possible scores range from 0-10, where lower scores indicate better outcome.
Change in pain scores as measured by Likert Scale Questionnaire | Baseline (before surgery in the pre-operative setting -Day 0), the day of ureter stent removal (Post-operative day 5 through 10)
  Associated pain burden will be measured using standardized Likert Scale Questionnaire. Possible scores range from 0-10, where lower scores indicate better outcome.
  For those patients in the SPIRIX arm, they will be asked to complete the Likert Scale Questionnaire approximately 30 minutes after taking each SPIRIX dose.

SECONDARY OUTCOMES:
Number of unplanned clinical encounters | Post-operative setting -the day of ureter stent removal (Post-operative day 5 through 10)
  number of clinical encounters (i.e. telephone calls, MyChart messages, emergency room visits, hospital readmissions) related to ureter stent discomfort will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Johnson, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearle MS. Medical therapy for urinary stone passage. Lancet. 2006 Sep 30;368(9542):1138-9. doi: 10.1016/S0140-6736(06)69452-X. No abstract available. PMID 17011928
- [Background] Bensalah K, Tuncel A, Gupta A, Raman JD, Pearle MS, Lotan Y. Determinants of quality of life for patients with kidney stones. J Urol. 2008 Jun;179(6):2238-43; discussion 2243. doi: 10.1016/j.juro.2008.01.116. Epub 2008 Apr 18. PMID 18423704
- [Background] Saigal CS, Joyce G, Timilsina AR; Urologic Diseases in America Project. Direct and indirect costs of nephrolithiasis in an employed population: opportunity for disease management? Kidney Int. 2005 Oct;68(4):1808-14. doi: 10.1111/j.1523-1755.2005.00599.x. PMID 16164658
- [Background] Shoag J, Halpern J, Goldfarb DS, Eisner BH. Risk of chronic and end stage kidney disease in patients with nephrolithiasis. J Urol. 2014 Nov;192(5):1440-5. doi: 10.1016/j.juro.2014.05.117. Epub 2014 Jun 11. PMID 24929140
- [Background] Alexander RT, Hemmelgarn BR, Wiebe N, Bello A, Morgan C, Samuel S, Klarenbach SW, Curhan GC, Tonelli M; Alberta Kidney Disease Network. Kidney stones and kidney function loss: a cohort study. BMJ. 2012 Aug 29;345:e5287. doi: 10.1136/bmj.e5287. PMID 22936784
- [Background] Ljunghall S, Danielson BG. A prospective study of renal stone recurrences. Br J Urol. 1984 Apr;56(2):122-4. doi: 10.1111/j.1464-410x.1984.tb05346.x. PMID 6498430
- [Background] Uribarri J, Oh MS, Carroll HJ. The first kidney stone. Ann Intern Med. 1989 Dec 15;111(12):1006-9. doi: 10.7326/0003-4819-111-12-1006. PMID 2688503
- [Background] Vadivelu N, Gowda AM, Urman RD, Jolly S, Kodumudi V, Maria M, Taylor R Jr, Pergolizzi JV Jr. Ketorolac tromethamine - routes and clinical implications. Pain Pract. 2015 Feb;15(2):175-93. doi: 10.1111/papr.12198. Epub 2014 Apr 16. PMID 24738596
- [Background] Singla N, Singla S, Minkowitz HS, Moodie J, Brown C. Intranasal ketorolac for acute postoperative pain. Curr Med Res Opin. 2010 Aug;26(8):1915-23. doi: 10.1185/03007995.2010.495564. PMID 20557145
- [Background] Johnson BA, Sorokin I, Antonelli J, Pearle M. Efficacy of Intramuscular Ketorolac for Preventing Renal Colic Post Stent Removal: Randomized Controlled Trial. J Urol. 2022 Sep;208(3):650-657. doi: 10.1097/JU.0000000000002750. Epub 2022 Jun 2. PMID 35653577
- [Background] Harper JD, Desai AC, Antonelli JA, Tasian GE, Ziemba JB, Al-Khalidi HR, Lai HH, Maalouf NM, Reese PP, Wessells HB, Kirkali Z, Scales CD Jr; NIDDK Urinary Stone Disease Research Network (USDRN). Quality of life impact and recovery after ureteroscopy and stent insertion: insights from daily surveys in STENTS. BMC Urol. 2022 Apr 6;22(1):53. doi: 10.1186/s12894-022-01004-9. PMID 35387623
- [Background] Allam CL, Aden JK, Reed AM. The Role of Routine Ureteral Stenting Following Uncomplicated Ureteroscopic Treatment for Upper Ureteral and Renal Stones: A Randomized Control Trial. J Endourol. 2023 Mar;37(3):257-263. doi: 10.1089/end.2022.0386. Epub 2023 Jan 9. PMID 36401514